CLINICAL TRIAL: NCT03795207
Title: A Randomized Phase II Trial of Stereotactic Body Radiation Therapy (SBRT) With or Without Durvalumab (MEDI4736) in Oligometastatic Recurrent Hormone Sensitive Prostate Cancer Patients
Brief Title: Prostate Cancer With OligometaSTatic Relapse: Combining Stereotactic Ablative Radiotherapy and Durvalumab (MEDI4736)
Acronym: POSTCARD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICO-N-2017-08
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Node; Prostate; Bone Metastases; Prostate Cancer Patients
Keywords: Node; Prostate; Bone Metastases; Prostate cancer patients; SBRT (Stereotactic body radiation therapy); Durvalumab; TEP-FCH; TEP-PSMA
MeSH Terms: interventions — Radiosurgery; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm SBRT + DURVALUMAB (Experimental): Radiation (SBRT) + Immunotherapy treatment (Durvalumab)
  64 patients will be enrolled in this arm
  Durvalumab, will be started one month prior to SBRT and then given for a total of 12 months.
  Patient will receive one injection per months (1500 mg/cycle)
  SBRT will be started one month after Durvalumab and patients will receive 3 fractions of radiation
  Interventions: Combination Product: SBRT + Durvalumab
- Arm SBRT (Active Comparator): Radiation (SBRT)
  32 patients will be enrolled in this arm
  Patients will receive only 3 fractions of radiation
  Interventions: Radiation: SBRT

INTERVENTIONS:
Combination Product: SBRT + Durvalumab — Durvalumab, MEDI4736, is a immunotherapy,
  SBRT (stereotactic body radiotherapy) is a procedure that uses high doses of radiation delivered to a precise target. By using special positioning and implanted markers in the body, radiologists are able to deliver a much higher dose of radiation to a cancer than traditional radiation therapy
  Arms: Arm SBRT + DURVALUMAB
Radiation: SBRT — SBRT (stereotactic body radiotherapy) is a procedure that uses high doses of radiation delivered to a precise target. By using special positioning and implanted markers in the body, radiologists are able to deliver a much higher dose of radiation to a cancer than traditional radiation therapy
  Arms: Arm SBRT

SUMMARY:
As in other solid tumours, increasing evidence indicates that patients diagnosed with a limited number of prostate cancer metastases, so-called oligometastases, have a better prognosis compared with patients with extensive metastatic disease.

Survival of patients with three or fewer metastases was superior compared with patients with more than three lesions.

The introduction of novel imaging modalities such as Fluorocholine (FCH), Fuciclovine or Ga-PSMA PET CT has increased the detection of oligometastatic prostate cancer (PCa) recurrence, potentially justifying the use of a metastasis-directed therapy with radiotherapy (RT).

Based on several studies, SBRT is now considered as a strongly validated option in oligometastatic prostate cancer.

It is increasingly understood that cancers are recognized by the immune system, and, under some circumstances, the immune system may control or even eliminate tumors.

Programmed death-ligand 1 (PD-L1) is transmembrane protein that has been speculated to play a major role in suppressing the immune system during particular events.

PD-L1 is expressed in a broad range of cancers. Based on these findings, an anti-PD-L1 antibody could be used therapeutically to enhance antitumor immune responses in patients with cancer.

Experimental data from multiple cancer models have provided cumulative evidence of an interaction of ionizing radiation with the systemic antitumor immunity and this has created several opportunities in the field.

The oligometastatic setting appears to be the most relevant clinical situation to evaluate the immune response generated by radiotherapy and immune modifiers in patients with an intact immune system. The hypothesize is that Durvalumab will enhance immune response following SBRT targeting oligometastatic lesions. In this randomized 2:1 phase II trial of Stereotactic Body Radiation Therapy with or without durvalumab in oligometastatic hormone sensitive prostate cancer patients, Durvalumab will be started one month prior to SBRT to be able to evaluate PSA and immune response to the drug. It will be combined with SBRT and then given adjuvantly for a total of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the patient prior to performing any protocol-related procedures, including screening evaluations
2. Age > or = 18 years at time of study entry
3. Histologically proven diagnosis of prostate cancer (PCa)
4. PCa patients with a biochemical recurrence "Rising PSA" following treatment with curative intent (radical prostatectomy, primary radiotherapy or a combination of both) as defined by the EAU guidelines.
5. A maximum of 5 bone or lymph node metastases, seen only on FCH-PET CT or Ga-PSMA PET CT, not seen on conventional imaging assessments (bone scan or thorax, abdomen and pelvis CT scan).
6. WHO performance state 0-1
7. Controlled primary tumor. In case the PSA > 0,2 ng/ml in the postoperative setting patients are eligible if a multiparametic MRI or PET scan of the prostate bed rules out a local relapse.

   Patients after primary radiotherapy should undergo MRI of the prostate according to the European Society of Urogenital Radiology (ESUR) guidelines to rule out local relapse. In case of a suspicious lesion, a biopsy should confirm local recurrence and patients should be referred for local salvage prostatectomy when distant metastases are ruled out. If MRI rules out local relapse, patients are eligible.
8. If ADT has been previously administered to the patient, a minimum of 12 months must have elapsed between the predicted duration of the last injection and inclusion of the patient in the study. For this category of patients, serum testosterone has to be higher than 8.5 nmol/l prior to inclusion.
9. Adequate normal organ and marrow function as defined below:

   * Haemoglobin ≥9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1.5 x 103 /L (≥ 1500 per mm3)
   * Platelet count ≥ 75 x 109/L (≥75,000 per mm3)
   * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysishaemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
   * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
   * Measured creatinine clearance (CL) ≥ 40 ml/min or Calculated creatinine CL ≥ 40 ml/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance: Creatinine CL (ml/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)
10. Body weight > 30kg
11. Life expectancy of > 24 months.
12. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
13. Social insurance

Exclusion Criteria:

1. Serum testosterone level < 8.5 nmol/ml
2. Vertebral metastases with a minimum distance inferior to 5 mm between GTV (gross tumor volume) and spinal cord
3. Visceral metastases
4. Bone metastases seen on bone scan
5. Lymph nodes greater than 20 mm
6. PSA doubling time less than 6 months
7. Spinal cord compression
8. Any unresolved toxicity NCI CTCAE (v4.03) Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
9. PSA rise while on active treatment (LHRH-agonist, LHRH-antagonist, anti-androgen, maximal androgen blockade, oestrogen)
10. Lung, Brain, Liver or other visceral metastases
11. Relapsed primary tumor
12. Perihilar lymphnode metastases
13. Previous irradiation of the oligometastatic site using a dose > 20 Gy less than 5 years ago.
14. Previous treatment with a cytotoxic agent for PCa
15. Treatment during the past month with products known to influence PSA levels (e.g. fluconazole, finasteride, corticosteroids...)
16. Particimmunotherapyation in another clinical study with an investigational product during the last 4 weeks
17. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
18. Any prior immune therapy (CTLA-4, PD1 (Programmed cell death )1 or PD-L1 inhibitor, including durvalumab)
19. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
20. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug
21. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of Durvalumab.
22. History of allogenic organ transplantation.
23. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    * Patients with celiac disease controlled by diet alone
24. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement
25. History of another primary malignancy except for

    * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of immunotherapy and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
26. History of leptomeningeal carcinomatosis
27. History of active primary immunodeficiency
28. Active infection including tuberculosis, hepatitis B (known positive HBV (hepatitis B virus) surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV (hepatitis B virus) infection (defined as the presence of hepatitis B core antibody [anti-HBc (hepatitis B core antigen)] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
29. Receipt of live attenuated vaccine within 30 days prior to the first dose of immunotherapy. Note: Patients, if enrolled, should not receive live vaccine whilst receiving immunotherapy and up to 30 days after the last dose of immunotherapy.
30. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
31. Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
32. Male patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2027-12-27 (Estimated)

PRIMARY OUTCOMES:
Two-years Progression-free survival | 54 months
  The primary outcome will be progression-free survival, defined as the time from randomization until a biochemical-clinical failure

SECONDARY OUTCOMES:
Health-related quality of life | through study completion, an average of 7.5 year
  Health-related quality of life will be evaluated using EORTC QLQ-PR25 instruments.Total score is reported
Health-related quality of life | through study completion, an average of 7.5 year
  Health-related quality of life will be evaluated using self-administered EORTC QLQ-C30 questionnaire. Total score is reported
Androgen deprivation therapy free survival | through study completion, an average of 7.5 year
  ADT will be started in both arms at time of polymetastatic disease, local progression of metastases or symptoms.
Prostate cancer specific survival | through study completion, an average of 7.5 year
  Delay from randomization to death
Overall survival | through study completion, an average of 7.5 year
  Delay from randomization to death
Acute toxicity: Common toxicity criteria version 4.03 | through study completion, an average of 7.5 year
  Common toxicity criteria version 4.03
Late toxicity: Common toxicity criteria version 4.03 | through study completion, an average of 7.5 year
  Common toxicity criteria version 4.03
Time to resistance castration | through study completion, an average of 7.5 year
  serum testosterone measure

CONTACTS AND LOCATIONS:
Overall Officials: STEPHANE SUPIOT, Study Director — INSTITUT DE CANCEROLOGIE DE L'OUEST
Locations (9):
- France (9):
  - Institut Bergonie, Bordeaux
  - CHRU de Brest, Brest
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Chbs Lorient, Lorient
  - Centre Léon Bérard, Lyon
  - Institut de Cancérologie de Montpellier, Montpellier
  - Hospices Civils de Lyon, Pierre-Bénite
  - ICO, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No